CLINICAL TRIAL: NCT01992107
Title: A Phase III, Stratified, Randomized, Double-Blind, Multicenter, Non-Inferiority Study to Evaluate Safety and Immunogenicity of Cell-Based Quadrivalent Subunit Influenza Virus Vaccine and Cell-Based Trivalent Subunit Influenza Virus Vaccines in Subjects Ages ≥4 Years to < 18 Years
Brief Title: Safety and Immunogenicity of Three Influenza Vaccines in Children Aged 4 Years Old to Less Than 18 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V130_03
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-11

CONDITIONS: Influenza
Keywords: Influenza; Influenza vaccine; Novartis; children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- QIVc (≥4 to <18 years) (Experimental): Subjects received one or two doses of QIVc-Quadrivalent Cell-based Influenza Vaccine recommended for 2013-2014 season
  Interventions: Biological: QIVc
- TIV1c (≥4 to <18 years) (Active Comparator): Subjects received one or two doses of TIV1c (Trivalent Inactivated Cell-based Influenza Vaccine containing one strain from B lineage ("B1" strain) recommended for 2013-2014 season
  Interventions: Biological: TIV1c
- TIV2c (≥4 to <18 years) (Active Comparator): Subjects received one or two doses of TIV2c (Trivalent Inactivated Cell-based Influenza Vaccine containing B strain from the alternate lineage ("B2" strain) recommended for 2013-2014
  Interventions: Biological: TIV2c

INTERVENTIONS:
Biological: QIVc — Novartis Investigational Quadrivalent Vaccine
  Arms: QIVc (≥4 to <18 years)
Biological: TIV1c — Licensed Influenza Vaccine
  Arms: TIV1c (≥4 to <18 years)
Biological: TIV2c — Novartis Investigational Vaccine
  Arms: TIV2c (≥4 to <18 years)

SUMMARY:
Evaluate safety and immunogenicity of three influenza vaccines in children ages greater than 4 years old to less than 18 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 4 years to less than 18 years of age.
2. Individual who had a parent or guardian who could give written informed consent after understanding the nature of the study and comply with study procedures and were available for follow-up.
3. If the individual was of an age where, according to local regulations, informed assent is required, that individual had provided assent to participate in the study.

Exclusion Criteria:

1. Individuals recently vaccinated against influenza
2. Subjects with contraindications to receive influenza vaccine

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2333 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (76):
- United States (76):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Harrisburg, Arkansas
  - Jonesboro, Arkansas
  - Anaheim, California
  - Downey, California
  - Garden Grove, California
  - Modesto, California
  - Paramount, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Santa Rosa, California
  - West Covina, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Thornton, Colorado
  - Boca Raton, Florida
  - Lake Mary, Florida
  - Melbourne, Florida
  - Miami Beach, Florida
  - Opa-locka, Florida
  - Pinellas Park, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Woodstock, Georgia
  - Boise, Idaho
  - Peoria, Illinois
  - Mishawaka, Indiana
  - Council Bluffs, Iowa
  - Newton, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Metairie, Louisiana
  - Kansas City, Missouri
  - St Louis, Missouri
  - Bellevue, Nebraska
  - Fremont, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Binghamton, New York
  - Wilmington, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Kettering, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Erie, Pennsylvania
  - Hermitage, Pennsylvania
  - Sellersville, Pennsylvania
  - Upper Saint Clair, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Bristol, Tennessee
  - Jefferson City, Tennessee
  - Lebanon, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Round Rock, Texas
  - San Angelo, Texas
  - San Antonio, Texas
  - Draper, Utah
  - Layton, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah
  - West Jordan, Utah
  - Burke, Virginia
  - Charlottesville, Virginia

REFERENCES:
- [Derived] Hartvickson R, Cruz M, Ervin J, Brandon D, Forleo-Neto E, Dagnew AF, Chandra R, Lindert K, Mateen AA. Non-inferiority of mammalian cell-derived quadrivalent subunit influenza virus vaccines compared to trivalent subunit influenza virus vaccines in healthy children: a phase III randomized, multicenter, double-blind clinical trial. Int J Infect Dis. 2015 Dec;41:65-72. doi: 10.1016/j.ijid.2015.11.004. Epub 2015 Nov 14. PMID 26585940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 90 centers in the United States (US)
Pre-assignment Details: All enrolled subjects were included in the trial
Groups:
- QIVc: Subjects received one or two doses of cell derived quadrivalent influenza vaccine (QIVc) recommended for 2013-2014 season
- TIV1c: Subjects received one or two doses of cell derived trivalent influenza vaccine TIV1c (H1N1, H3N2, B1) recommended for 2013-2014 season
- TIV2c: Subjects received one or two doses of cell derived trivalent influenza vaccine TIV2c that contains an alternate B strain compared to what is recommended for 2013-2014
Period: Overall Study
Arm/Group | QIVc | TIV1c | TIV2c
Started | 1159 | 593 | 581
Completed | 1091 | 560 | 545
Not Completed | 68 | 33 | 36
Not completed — Administrative reasons | 2 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 46 | 22 | 26
Not completed — noncompliance and were unavailable | 7 | 3 | 2
Not completed — Withdrawal by Subject | 13 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QIVc | TIV1c | TIV2c | Total
Number analyzed (Participants) | 1159 | 593 | 581 | 2333
Age, Continuous [Mean (Standard Deviation); unit: year] | 9.5 (3.8) | 9.5 (3.8) | 9.3 (3.7) | 9.5 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 556 | 284 | 284 | 1124
  Male | 603 | 309 | 297 | 1209

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titre (GMT) in Subjects After Receiving One or Two Doses of Either QIVc, TIV1c or TIV2c
Description: Immunogenicity of QIVc to comparator TIV1c (For A/H1N1, A/H3N2 and B1 strain, the comparison was between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison was between QIVc and TIV2c) was assessed in terms of GMT in subjects (Previously vaccinated and Not previously vaccinated) measured by hemagglutination inhibition (HI) assay, three weeks after last vaccination with one or two doses of either QIVc, TIV1c or TIV2c.
  Non-inferiority was established if the upper bound of the two-sided 95% confidence interval (CI) for the ratio of GMTs (GMT TIV1c or TIV2c /GMT QIVc) for HI antibody does not exceed the non-inferiority margin of 1.5.
Time Frame: Day 1,Three weeks post vaccination (Day 22 for previously vaccinated and Day 50 for Not previously vaccinated subjects)
Population: Analysis was done on Per Protocol (PP) Population i.e. all subjects in the Full Analysis Set (FAS) efficacy/immunogenicity population correctly received the vaccine, had no major protocol deviations leading to exclusion as defined prior to unblinding/analysis and are not excluded due to other reasons defined prior to unblinding or analysis
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- QIVc (≥4 to <18 Years): Subjects received one or two doses of cell derived quadrivalent influenza vaccine (QIVc) recommended for 2013-2014 season
- TIV1c (≥4 to <18 Years): Subjects received one or two doses of cell derived trivalent influenza vaccine TIV1c (H1N1, H3N2, B1) recommended for 2013-2014 season
- TIV2c (≥4 to <18 Years): Subjects received one or two doses of cell derived trivalent influenza vaccine TIV2c that contains an alternate B strain compared to what is recommended for 2013-2014
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593 | 581
Titers
  A/H1N1: Day 1 (N=1014, 510) | 96 [86 to 107] | 100 [86 to 116] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H1N1: Day 22/Day 50 (N=1014, 510) | 1090 [1027 to 1157] | 1125 [1034 to 1224] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: Day 1 (N=1013, 510) | 206 [188 to 225] | 196 [172 to 222] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: Day 22/Day 50 (N=1013, 510) | 738 [703 to 774] | 776 [725 to 831] | NA [NA to 0] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: Day 1 (N=1013, 510) | 26 [24 to 28] | 23 [21 to 26] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: Day 22/Day 50 (N=1013, 510) | 155 [146 to 165] | 154 [141 to 168] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B2: Day 1(N=1009, 501) | 23 [21 to 25] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 23 [21 to 26]
  B2: Day 22/Day 50 (N=1009, 501) | 185 [171 to 200] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 185 [166 to 207]
Statistical Analysis 1: Comparison: QIVc (≥4 to <18 Years) vs TIV1c (≥4 to <18 Years); Non-inferiority of immune responses of QIVc to TIV1c, assessed in terms of ratios of GMT against influenza strain A/H1N1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the upper bound of the two-sided 95% confidence interval (CI) for the ratio of GMTs (GMT TIV1c/GMT QIVc) for HI antibody does not exceed the non-inferiority margin of 1.5; ANCOVA; Ratios of GMT (Day 22/Day 50) = 1.03, 95% CI 2-sided [0.93 to 1.14]
Statistical Analysis 2: Comparison: QIVc (≥4 to <18 Years) vs TIV1c (≥4 to <18 Years); Non-inferiority of immune responses of QIVc to TIV1c, assessed in terms of ratios of GMT against influenza strain A/H3N2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratios of GMT (Day 22/Day 50) = 1.05, 95% CI 2-sided [0.97 to 1.14]
Statistical Analysis 3: Comparison: QIVc (≥4 to <18 Years) vs TIV1c (≥4 to <18 Years); Non-inferiority of immune responses of QIVc to TIV1c, assessed in terms of ratios of GMT against influenza strain B1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratios of GMT (Day 22/Day 50) = 0.99, 95% CI 2-sided [0.89 to 1.1]
Statistical Analysis 4: Comparison: QIVc (≥4 to <18 Years) vs TIV2c (≥4 to <18 Years); Non-inferiority of immune responses of QIVc to TIV2c, assessed in terms of ratios of GMT against influenza strain B2; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the upper bound of the two-sided 95% confidence interval (CI) for the ratio of GMTs (GMT TIV2c/GMT QIVc) for HI antibody does not exceed the non-inferiority margin of 1.5; ANCOVA; Ratios of GMT (Day 22/Day 50) = 1, 95% CI 2-sided [0.87 to 1.14]

2. Primary Outcome: Percentages of Subjects Achieving Seroconversion After One or Two Doses of Either QIVc, TIV1c or TIV2c
Description: Immunogenicity of QIVc to comparator TIVc (For A/H1N1, A/H3N2 and B1 strain, the comparison was between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison was between QIVc and TIV2c) was assessed in terms of number (%) of subjects (Previously vaccinated and Not previously vaccinated) showing seroconversion or significant increase (at least a 4-fold increase in HI titer in subjects seropositive at baseline [i.e., HI titer ≥1:10 at Day 1] ) in HI antibody titers, three weeks after last vaccination with one or two doses of either QIVc, TIV1c or TIV2c Seroconversion was defined in subjects seronegative at baseline (i.e., HI titer <1:10 at Day 1) as postvaccination HI titer ≥1:40, and defined in subjects seropositive at baseline (i.e., HI titer ≥1:10 at Day 1) as a minimum of a 4-fold increase in post-vaccination HI titer.
Time Frame: Three weeks post vaccination (Day 22 for previously vaccinated and Day 50 for Not previously vaccinated subjects)
Population: Analysis was done on PP population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593 | 581
percentages of subjects
  A/H1N1: Day 22/Day 50 (N=1014,510) | 72 [69 to 75] | 75 [70 to 78] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: Day 22/Day 50 (N=1013, 510) | 47 [44 to 50] | 51 [46 to 55] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: Day 22/Day 50 (N=1013,510) | 66 [63 to 69] | 66 [62 to 70] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B2: Day 22/Day 50 (N=1009,501) | 73 [70 to 76] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 71 [67 to 75]
Statistical Analysis 1: Comparison: QIVc (≥4 to <18 Years) vs TIV1c (≥4 to <18 Years); Non-inferiority of immune responses of QIVc to TIV1c in terms of differences in seroconversion rates against influenza strain A/H1N1; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the upper bound of the two-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV1c - % seroconversion QIVc) for HI antibody does not exceed the margin of 10%; ANCOVA; Difference b/w SC rates (Day 22/Day 50) = 2, 95% CI 2-sided [-2.5 to 6.9]
Statistical Analysis 2: Comparison: QIVc (≥4 to <18 Years) vs TIV1c (≥4 to <18 Years); Non-inferiority of immune responses of QIVc to TIV1c in terms of differences in seroconversion rates against influenza strain A/H3N2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Difference b/w SC rates (Day 22/Day 50) = 4, 95% CI 2-sided [-1.4 to 9.2]
Statistical Analysis 3: Comparison: QIVc (≥4 to <18 Years) vs TIV1c (≥4 to <18 Years); Non-inferiority of immune responses of QIVc to TIV1c in terms of differences in seroconversion rates against influenza strain B1; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Difference b/w SC rates (Day 22/Day 50) = 0, 95% CI 2-sided [-5.5 to 4.5]
Statistical Analysis 4: Comparison: QIVc (≥4 to <18 Years) vs TIV2c (≥4 to <18 Years); Non-inferiority of immune responses of QIVc to TIV2c in terms of differences in seroconversion rates against influenza strain B2; Test type: Non-Inferiority or Equivalence — Non-inferiority was established if the upper bound of the two-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV2c - % seroconversion QIVc) for HI antibody does not exceed the margin of 10%; ANCOVA; Difference b/w SC rates (Day 22/Day 50) = -2, 95% CI 2-sided [-6.5 to 3.2]

3. Secondary Outcome: Percentages of Subjects Achieving Seroconversion After One or Two Doses of Either QIVc, TIV1c or TIV2c in ≥4 to <18 Years
Description: Immunogenicity was assessed in terms of number (%) of subjects (Previously vaccinated and Not previously vaccinated) showing seroconversion or significant increase in HI antibody titers, three weeks after last vaccination with one or two doses of either QIVc, TIV1c or TIV2c For A/H1N1, A/H3N2 and B1 strain, the comparison was between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison was between QIVc and TIV2c Seroconversion was defined in subjects seronegative at baseline (i.e., HI titer <1:10 at Day 1) as postvaccination HI titer ≥1:40, and defined in subjects seropositive at baseline (i.e., HI titer ≥1:10 at Day 1) as a minimum of a 4-fold increase in post-vaccination HI titer.
  The Center for Biologics Evaluation, Research, and Review (CBER) criterion for an adult population is that the lower bound of the two-sided 95% CI for the percentage of subjects achieving seroconversion for HI antibody should meet or exceed 40%
Time Frame: Three weeks post vaccination (Day 22 for previously vaccinated and Day 50 for Not previously vaccinated subjects)
Population: Analysis was done on Full Analysis Set (FAS) immunogenicity set i.e. all subjects in the enrolled set who received ▫ Received at least one study vaccination and provided immunogenicity data at day 1 and day 22 (day 50 for not previously vaccinated subjects)
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593 | 581
percentages of subjects
  A/H1N1: Day 22 or Day 50 (N=1113,566) | 73 [70 to 76] | 74 [70 to 77] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: Day 22 or Day 50 (N=1112,566) | 47 [44 to 50] | 51 [47 to 55] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: Day 22 or Day 50 (N=1112,566) | 67 [64 to 70] | 66 [61 to 69] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B2: Day 22 or Day 50 (N=1108,556) | 73 [70 to 76] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 72 [68 to 76]

4. Secondary Outcome: Percentages of Subjects Achieving HI Titer ≥1:40 After One or Two Doses of Either QIVc, TIV1c or TIV2c in ≥4 to <18 Years
Description: Immunogenicity was assessed in terms of number (%) of subjects (Previously vaccinated and Not previously vaccinated) showing HI titer ≥1:40, three weeks after last vaccination with one or two doses of either QIVc, TIV1c or TIV2c For A/H1N1, A/H3N2 and B1 strain, the comparison was between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison was between QIVc and TIV2c.
  The CBER criterion for adult population was that the lower bound of the two-sided 95% CI for the percentage of subjects achieving an HI antibody titer ≥1:40 should meet or exceed 70%
Time Frame: Day 1, Three weeks post vaccination (Day 22 for previously vaccinated and Day 50 for Not previously vaccinated subjects)
Population: Analysis was done on FAS immunogenicity set (FAS) i.e. all subjects in the enrolled set who received at least one study vaccination and provided immunogenicity data at day 22 (day 50 for not previously vaccinated subjects)
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593 | 581
percentages of subjects
  A/H1N1: Day 1(N=1113,566) | 76 [73 to 78] | 79 [75 to 82] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H1N1: Day 22 or Day 50(N=1113,566) | 99 [98 to 100] | 99 [98 to 100] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: Day 1(N=1112,566) | 90 [88 to 91] | 89 [86 to 92] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: Day 22 or Day 50(N=1112,566) | 100 [99 to 100] | 99 [98 to 100] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: Day 1(N=1112,566) | 49 [46 to 52] | 45 [41 to 49] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: Day 22 or Day 50(N=1112,566) | 92 [91 to 94] | 93 [90 to 95] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B2: Day 1(N=1108,556) | 46 [43 to 49] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 47 [43 to 51]
  B2: Day 22 or Day 50(N=1108,556) | 91 [89 to 93] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 91 [88 to 93]

5. Secondary Outcome: Percentages of Subjects Achieving Seroconversion After One or Two Doses of Either QIVc, TIV1c or TIV2c in ≥4 to <18 Years
Description: Immunogenicity was assessed in terms of number (%) of subjects (Previously vaccinated and Not previously vaccinated) showing seroconversion or significant increase in HI antibody titers, three weeks after last vaccination with one or two doses of either QIVc, TIV1c or TIV2c For A/H1N1, A/H3N2 and B1 strain, the comparison was between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison was between QIVc and TIV2c Seroconversion was defined in subjects seronegative at baseline (i.e., HI titer <1:10 at Day 1) as postvaccination HI titer ≥1:40, and defined in subjects seropositive at baseline (i.e., HI titer ≥1:10 at Day 1) as a minimum of a 4-fold increase in post-vaccination HI titer.
Time Frame: Three weeks post vaccination (Day 22 for previously vaccinated and Day 50 for Not previously vaccinated subjects)
Population: Analysis was done on FAS immunogenicity set
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593 | 581
percentages of subjects
  A/H1N1: Day 22/Day 50(N=1113,566) | 73 [70 to 76] | 74 [70 to 77] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: Day 22/Day 50(N=1112,566) | 47 [44 to 50] | 51 [47 to 55] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: Day 22/Day 50(N=1112,566) | 67 [64 to 70] | 66 [61 to 69] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B2: Day 22/Day 50(N=1108,556) | 73 [70 to 76] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 72 [68 to 76]

6. Secondary Outcome: Percentages of Subjects Achieving HI Titer ≥1:40 After One or Two Doses of Either QIVc, TIV1c or TIV2c in ≥4 to <18 Years
Description: Immunogenicity was assessed in terms of number (%) of subjects (Previously vaccinated and Not previously vaccinated) showing HI titer ≥1:40, three weeks after last vaccination with one or two doses of either QIVc, TIV1c or TIV2c For A/H1N1, A/H3N2 and B1 strain, the comparison was between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison was between QIVc and TIV2c The Committee for Medicinal Products for Human Use (CHMP) criterion for an adult population was that the percentage of subjects achieving an HI titer ≥1:40 is >70%
Time Frame: as for outcome 4
Population: Analysis was done on FAS immunogenicity set
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593 | 581
percentages of subjects
  A/H1N1: Day 1(N=1113,566) | 76 [73 to 78] | 79 [75 to 82] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H1N1: Day 22/Day 50(N=1113,566) | 99 [98 to 100] | 99 [98 to 100] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: Day 1(N=1112,566) | 90 [88 to 91] | 89 [86 to 92] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: Day 22/Day 50(N=1112,566) | 100 [99 to 100] | 99 [98 to 100] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: Day 1(N=1112,566) | 49 [46 to 52] | 45 [41 to 49] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: Day 22/Day 50(N=1112,566) | 92 [91 to 94] | 93 [90 to 95] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B2: Day 1(N=1108,556) | 46 [43 to 49] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 47 [43 to 51]
  B2: Day 22/Day 50(N=1108,556) | 91 [89 to 93] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 91 [88 to 93]

7. Secondary Outcome: Geometric Mean Ratios (GMR) in Subjects After One or Two Doses of Either QIVc, TIV1c or TIV2c in ≥4 to <18 Years Age
Description: Immunogenicity was measured in subjects (Previously vaccinated and Not previously vaccinated) as the geometric mean ratio (GMR). The ratio of postvaccination to prevaccination HI GMTs, three weeks after last vaccination with one or two doses of either QIVc, TIV1c or TIV2c .For A/H1N1, A/H3N2 and B1 strain, the comparison was between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison was between QIVc and TIV2c The CHMP criterion for GMR in adult population is >2.5
Time Frame: Three weeks post vaccination (Day 22 for previously vaccinated and Day 50 for Not previously vaccinated subjects)
Population: Analysis was done on FAS immunogenicity set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593 | 581
Ratios
  A/H1N1: TIV1c/QIVc [Day 22 (Day 50)/Day1] | 11 [10 to 13] | 12 [10 to 13] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  A/H3N2: TIV1c/QIVc [Day 22 (Day 50)/Day1] | 3.65 [3.4 to 3.91] | 3.97 [3.59 to 4.38] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B1: TIV1c/QIVc [Day 22 (Day 50)/Day1] | 6.15 [5.72 to 6.61] | 6.24 [5.64 to 6.91] | NA [NA to NA] — Participants in the TIV2c Arm/Group were not vaccinated with the H1N1, H3N2 and B1 strains
  B2: TIV2c/QIVc [Day 22 (Day 50)/Day1] | 8.17 [7.5 to 8.89] | NA [NA to NA] — Participants in the TIV1c Arm/Group were not vaccinated with the B2 strain | 8.45 [7.5 to 9.53]

8. Secondary Outcome: GMT in Subjects After Receiving One or Two Doses of Either QIVc, TIV1c Against B2 Strain
Description: Immunogenicity of QIVc to comparator TIV1c was assessed in terms of GMT in subjects (Previously vaccinated and Not previously vaccinated) measured by HI assay, three weeks after last vaccination with one or two doses of either QIVc or TIV1c.
  Superiority was established if the upper bound of the two-sided 95% CI for the ratio of GMTs (GMT TIV1c /GMT QIVc) for HI antibody did not exceed the superiority margin of 1
Time Frame: as for outcome 4
Population: Analysis was done on FAS population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593
Titers
  Day1(N=1108,563) | 22 [20 to 24] | 21 [18 to 23]
  Day 22/Day 50(N=1108,563) | 176 [164 to 189] | 45 [41 to 49]
Statistical Analysis 1: Comparison: QIVc (≥4 to <18 Years) vs TIV1c (≥4 to <18 Years); Superiority of immune responses of QIVc to TIV1c in terms of ratios of GMT against influenza strain B2.The upper bound of the two-sided 95% CI for the ratio of GMTs (GMT TIV1c/GMTQIVc) for HI antibody should not exceed the superiority margin of 1 met; Test type: Superiority or Other; Ratios of GMT (Day 22/Day 50) = 0.25, 95% CI 2-sided [0.22 to 0.29]

9. Secondary Outcome: Percentages of Subjects Achieving Seroconversion Against B2 Strain After One or Two Doses of Either QIVc or TIV1c
Description: Immunogenicity of QIVc to comparator TIV1c in terms of number (%) of subjects (Previously vaccinated and Not previously vaccinated) showing seroconversion or significant increase in HI antibody titers, against influenza strain B2, three weeks after last vaccination with QIVc or TIV1c.
  Superiority criterion was established if the upper bound of the two-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV1c - % seroconversion QIVc) for HI antibody does not exceed the margin of 0 points
Time Frame: Three weeks post vaccination (Day 22 for previously vaccinated and Day 50 for Not previously vaccinated subjects)
Population: Analysis was done on FAS population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593
percentages of subjects | 73 [70 to 76] | 26 [23 to 30]
Statistical Analysis 1: Comparison: QIVc (≥4 to <18 Years) vs TIV1c (≥4 to <18 Years); Superiority of immune responses of QIVc to TIV1c in terms of seroconversion rates against influenza strain B2.The upper bound of the 2-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV1c - %seroconversion QIVc) for HI antibody should not exceed the margin of 0 points met; Test type: Superiority or Other; Difference b/w SC rates(Day 22/Day 50) = -47, 95% CI 2-sided [-51.1 to -42.1]

10. Secondary Outcome: GMT in Subjects After Receiving One or Two Doses of Either QIVc,TIV2c Against B1 Strain
Description: Immunogenicity of QIVc to comparator TIV2c was assessed in terms of GMT in subjects (Previously vaccinated and Not previously vaccinated) measured by HI assay, three weeks after last vaccination with one or two doses of either QIVc or TIV2c.
  Superiority was established if the upper bound of the two-sided 95% CI for the ratio of GMTs (GMT TIV2c /GMT QIVc) for HI antibody does not exceed the superiority margin of 1
Time Frame: as for outcome 4
Population: Analysis was done on FAS population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | QIVc (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 581
Titers
  Day1(N=1112,557) | 25 [23 to 27] | 24 [22 to 27]
  Day 22/Day 50(N=1112,557) | 154 [145 to 163] | 59 [54 to 64]
Statistical Analysis 1: Comparison: QIVc (≥4 to <18 Years) vs TIV2c (≥4 to <18 Years); Superiority of immune responses of QIVc to TIV2c in terms of ratios of GMT against influenza strain B1.The upper bound of the 2-sided 95% CI for the ratio of GMTs (GMT TIV2c /GMTQIVc) for HI antibody should not exceed the superiority margin of 1 met; Test type: Superiority or Other; Ratios of GMT (Day 22/Day 50) = 0.38, 95% CI 2-sided [0.35 to 0.42]

11. Secondary Outcome: Percentages of Subjects Achieving Seroconversion After One or Two Doses of Either QIVc or TIV2c
Description: Immunogenicity of QIVc to comparator TIV2c in terms of number (%) of subjects (Previously vaccinated and Not previously vaccinated) showing seroconversion or significant increase in HI antibody titers, against influenza strain B1, three weeks after last vaccination with QIVc or TIV2c.
  Superiority was established if the upper bound of the two-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV2c - % seroconversion QIVc) for HI antibody does not exceed the margin of 0 points
Time Frame: Three weeks post vaccination (Day 22 for previously vaccinated and Day 50 for Not previously vaccinated subjects)
Population: Analysis was done on FAS population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | QIVc (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 581
percentages of subjects | 67 [64 to 70] | 33 [29 to 37]
Statistical Analysis 1: Comparison: QIVc (≥4 to <18 Years) vs TIV2c (≥4 to <18 Years); Superiority of immune responses of QIVc to TIV2c in terms of seroconversion rates against influenza strain B1.The upper bound of the 2-sided 95% CI for the difference between seroconversion rates (% seroconversion TIV1c or TIV2c - %seroconversion QIVc) for HI antibody should not exceed the margin of 0 points met; Test type: Superiority or Other; Difference b/w SC rates(Day 22/Day 50) = -34, 95% CI 2-sided [-38.8 to -29.3]

12. Secondary Outcome: Number of Subjects Reporting Solicited Adverse Events (AEs) After One or Two Doses of Either QIVc, TIV1c or TIV2c by Age Sub-strata
Description: Safety was assessed in terms of number of subjects (Previously vaccinated and Not previously vaccinated) reporting solicited local and systemic reactions, day 1 to 7 after last vaccination with one or two doses of either QIVc, TIV1c or TIV2c.For A/H1N1, A/H3N2 and B1 strain, the comparison was between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison is between QIVc and TIV2c.
Time Frame: Day 1 to 7 after last vaccination
Population: Analysis was done on solicited safety data set i.e. all subjects in the exposed set with solicited adverse event data
Measure: Number; unit: Subjects
Groups:
- QIVc _First Vaccine (≥4 to <6 Years); QIVc _Second Vaccine (≥4 to <6 Years); QIVc _First Vaccine (≥6 to <9 Years); QIVc _Second Vaccine (≥6 to <9 Years): Subjects received one or two doses of cell derived quadrivalent influenza vaccine (QIVc) recommended for 2013-2014 season
- TIV1c_First Vaccine (≥4 to <6 Years); TIV1c_Second Vaccine (≥4 to <6 Years); TIV1c_Second Vaccine (≥6 to <9 Years): Subjects received one or two doses of cell derived trivalent influenza vaccine TIV1c (H1N1, H3N2, B1) recommended for 2013-2014 season
- TIV2c _First Vaccine (≥4 to <6 Years); TIV2c _Second Vaccine (≥4 to <6 Years); TIV2c _First Vaccine (≥6 to <9 Years); TIV2c _Second Vaccine (≥6 to <9 Years): Subjects received one or two doses of cell derived trivalent influenza vaccine TIV2c that contains an alternate B strain compared to what is recommended for 2013-2014
- TIV1c_First Vaccine (≥6 to <9 Years): Subjects received one or two doses of cell derived trivalent influenza vaccine TIV1c (H1N1, H3N2,B1) recommended for 2013-2014 season
- QIVc (≥9 to <18 Years): Subjects received one dose of cell derived quadrivalent influenza vaccine (QIVc) recommended for 2013-2014 season
- TIV1c (≥9 to <18 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV1c (H1N1, H3N2, B1) recommended for 2013-2014 season
- TIV2c (≥9 to <18 Years): Subjects received one dose of cell derived trivalent influenza vaccine TIV2c that contains an alternate B strain compared to what is recommended for 2013-2014
Arm/Group | QIVc _First Vaccine (≥4 to <6 Years) | TIV1c_First Vaccine (≥4 to <6 Years) | TIV2c _First Vaccine (≥4 to <6 Years) | QIVc _Second Vaccine (≥4 to <6 Years) | TIV1c_Second Vaccine (≥4 to <6 Years) | TIV2c _Second Vaccine (≥4 to <6 Years) | QIVc _First Vaccine (≥6 to <9 Years) | TIV1c_First Vaccine (≥6 to <9 Years) | TIV2c _First Vaccine (≥6 to <9 Years) | QIVc _Second Vaccine (≥6 to <9 Years) | TIV1c_Second Vaccine (≥6 to <9 Years) | TIV2c _Second Vaccine (≥6 to <9 Years) | QIVc (≥9 to <18 Years) | TIV1c (≥9 to <18 Years) | TIV2c (≥9 to <18 Years)
Number analyzed (Participants) | 182 | 91 | 93 | 98 | 39 | 47 | 372 | 185 | 186 | 205 | 112 | 116 | 579 | 294 | 282
Subjects
  Any local | 103 | 51 | 47 | 52 | 17 | 17 | 237 | 124 | 116 | 102 | 64 | 66 | 377 | 175 | 156
  Tenderness | 83 | 41 | 40 | 49 | 15 | 15 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ecchymosis | 16 | 10 | 7 | 6 | 3 | 2 | 35 | 17 | 14 | 9 | 9 | 7 | 24 | 16 | 13
  Erythema | 32 | 21 | 16 | 17 | 3 | 7 | 83 | 43 | 38 | 29 | 17 | 19 | 110 | 51 | 43
  Induration | 24 | 18 | 12 | 11 | 2 | 4 | 59 | 35 | 24 | 25 | 18 | 12 | 88 | 43 | 36
  Pain | 0 | 0 | 0 | 0 | 0 | 0 | 201 | 105 | 107 | 95 | 61 | 62 | 334 | 150 | 142
  Any systemic | 51 | 18 | 17 | 30 | 9 | 9 | 117 | 67 | 65 | 46 | 30 | 27 | 232 | 121 | 94
  Change of eating habits | 19 | 6 | 6 | 9 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sleepiness | 34 | 11 | 9 | 13 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills | 10 | 2 | 1 | 4 | 2 | 1 | 16 | 6 | 8 | 2 | 3 | 0 | 43 | 17 | 10
  Irritability | 29 | 9 | 9 | 15 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 9 | 10 | 7 | 6 | 4 | 55 | 24 | 21
  Myalgia | 0 | 0 | 0 | 0 | 0 | 0 | 43 | 26 | 19 | 18 | 11 | 11 | 94 | 50 | 41
  Arthralgia | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 10 | 7 | 6 | 5 | 4 | 36 | 19 | 22
  Headache | 0 | 0 | 0 | 0 | 0 | 0 | 52 | 24 | 23 | 9 | 8 | 7 | 127 | 68 | 50
  Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 47 | 26 | 33 | 18 | 12 | 10 | 104 | 46 | 44
  Vomiting | 8 | 2 | 2 | 3 | 0 | 0 | 12 | 6 | 6 | 7 | 2 | 1 | 10 | 4 | 5
  Diarrhea | 8 | 2 | 2 | 3 | 1 | 2 | 13 | 11 | 9 | 4 | 4 | 1 | 22 | 11 | 9
  Loss of appetite | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 10 | 15 | 6 | 9 | 8 | 51 | 25 | 25
  Body temperature(>=38C) | 7 | 4 | 3 | 4 | 1 | 0 | 16 | 5 | 4 | 6 | 2 | 2 | 7 | 8 | 4
  Analgesics and antipyretics-Preventive | 13 | 1 | 1 | 2 | 1 | 0 | 14 | 6 | 8 | 7 | 4 | 4 | 15 | 6 | 8
  Analgesics and antipyretics-Treatment | 12 | 4 | 3 | 2 | 2 | 1 | 27 | 13 | 10 | 15 | 4 | 10 | 24 | 20 | 14

13. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs After One or Two Doses of Either QIVc, TIV1c or TIV2c by Overall Age Group
Description: Safety was assessed in terms of number of subjects (Previously vaccinated and Not previously vaccinated) reporting unsolicited AEs (day 1 to 22 for Previously vaccinated and day 1 to day 50 for Not previously vaccinated subjects), serious adverse events (SAEs), medically attended AEs, AEs leading to withdrawal from the study, new onset of chronic diseases (NOCDs), and concomitant medications (day 1 to day 181 for Previously vaccinated and day 1 to day 210 for Not previously vaccinated subjects) after receiving one or two doses of either QIVc, TIV1c or TIV2c. For A/H1N1, A/H3N2 and B1 strain, the comparison is between QIVc and TIV1c and for B2 i.e. alternate B strain, the comparison was between QIVc and TIV2c.
Time Frame: Day 1 to 210 post vaccination
Population: Analysis was done on unsolicited safety data set i.e. all subjects in the exposed set with unsolicited adverse event data
Measure: Number; unit: Subjects
Arm/Group | QIVc (≥4 to <18 Years) | TIV1c (≥4 to <18 Years) | TIV2c (≥4 to <18 Years)
Number analyzed (Participants) | 1159 | 593 | 581
Subjects
  Any AE | 279 | 139 | 152
  Possibly/probably related AE | 56 | 34 | 31
  SAE | 6 | 7 | 2
  Possibly/probably related SAE | 0 | 0 | 0
  AE leading to study withdrawal | 0 | 1 | 0
  Medically attended AE | 310 | 156 | 153
  NOCD | 20 | 11 | 11
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period.
Description: Solicited AEs -collected from day 1 to day 7 after last vaccination, unsolicited AEs - collected from day 1 to day 22 for previously vaccinated subjects and day 1 to day 50 for not previously vaccinated subjects.SAEs were collected from day 1 to day 181 for previously vaccinated subjects and day 1 to day 210 for not previously vaccinated subjects
Groups:
- Total: Total number of Subjects
Arm/Group | QIVc | TIV1c | TIV2c | Total
Serious Adverse Events (participants affected / at risk) | 6/1149 | 7/579 | 2/570 | 15/2298
Other Adverse Events (participants affected / at risk) | 840/1149 | 417/579 | 392/570 | 1649/2298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QIVc (N=1149) | TIV1c (N=579) | TIV2c (N=570) | Total (N=2298)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0 | 0 | 1
ABSCESS OF EYELID (Infections and infestations) | 0 | 1 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 1 | 2
PERIORBITAL CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 1
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
HIPPOCAMPAL SCLEROSIS (Nervous system disorders) | 1 | 0 | 0 | 1
PARTIAL SEIZURES (Nervous system disorders) | 1 | 0 | 0 | 1
BIPOLAR DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 1
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 0 | 1 | 0 | 1
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 1
OPPOSITIONAL DEFIANT DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 1 | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1 | 0 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
HENOCH-SCHONLEIN PURPURA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QIVc (N=1149) | TIV1c (N=579) | TIV2c (N=570) | Total (N=2298)
DIARRHEA (Gastrointestinal disorders) | 66 | 33 | 28 | 127
NAUSEA (Gastrointestinal disorders) | 95 | 40 | 42 | 177
VOMITING (Gastrointestinal disorders) | 60 | 22 | 31 | 113
CHILLS (General disorders) | 73 | 29 | 21 | 123
FATIGUE (General disorders) | 165 | 82 | 82 | 329
INJECTION SITE ERYTHEMA (General disorders) | 244 | 121 | 110 | 475
INJECTION SITE HEMORRHAGE (General disorders) | 84 | 48 | 42 | 174
INJECTION SITE INDURATION (General disorders) | 188 | 105 | 78 | 371
INJECTION SITE PAIN (General disorders) | 664 | 324 | 315 | 1303
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 59 | 18 | 38 | 115
DECREASED APPETITE (Metabolism and nutrition disorders) | 92 | 43 | 45 | 180
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 63 | 35 | 33 | 131
MYALGIA (Musculoskeletal and connective tissue disorders) | 150 | 84 | 66 | 300
HEADACHE (Nervous system disorders) | 204 | 105 | 88 | 397
COUGH (Respiratory, thoracic and mediastinal disorders) | 45 | 34 | 24 | 103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.